CLINICAL TRIAL: NCT07197398
Title: Preoperative Data and the Spinal Spread of Local Anesthetic in Cesarean Section - a Retrospective Analysis of High Hyperbaric Bupivacaine Dose Cases.
Brief Title: Preoperative Data and the Spinal Spread of Local Anesthetic in Cesarean Section
Status: Recruiting | Type: Observational
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Bartosz Horosz, MD, Principal Investigator, Centre of Postgraduate Medical Education
Other Study IDs: 80/2025
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Spinal Anesthesia Evaluation; Cesarean Delivery
Keywords: spinal anesthesia; cesarean section; spinal dose; spinal block level
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parturients given spinal block with 12.5mg of hyperbaric bupivacaine: Hospital's electronic database will be searched in order to identify elective cases of cesarean sections performed under spinal anesthesia. After that, a manual review of each case will follow and only those where the dose of hyperbaric bupivacaine used for spinal block was 12.5mg will be chosen for further analysis. Anesthetic records of these cases will be retrieved and assessed for its quality, clarity and completeness. During the process of further analysis an anonymized data will be retrieved and moved to Excel file: demographic and pregnancy - related data of the parturient, spinal block - related data (technique and dynamic of the sensory blockade, maternal hemodynamic parameters) and neonatal data (birthweight). Special attention will be paid to assure that all data is accessible only for investigators and remain anonymous throughout the analysis process.
  Interventions: Other: Spinal block level analysis; Other: Data collection; Other: Sub-group analysis

INTERVENTIONS:
Other: Spinal block level analysis — Relation of pregnancy - related, maternal and neonatal data to the level of sensory blockade in the whole study group will be assessed. Only cases with 12.5mg of hyperbaric bupivacaine will be included.
Other: Data collection — Intervention is to retrieve and analyse anonymous perioperative data. After identification of eligible cases, statistical analysis will be performed
Other: Sub-group analysis — Relation of pregnancy - related, maternal and neonatal data to the level of sensory blockade in the sub-groups of different height (<165cm and >165cm) will also be performed.

SUMMARY:
This study is designed to assess possible relation between the anthropometric data of pregnant women at term, as well as their babies, and the maximal level of sensory blockade following spinal anesthesia for cesarean section. The debate regarding this relation is ongoing. Although there is some relevant data in favor of both lack and the presence of significant relation between these variables, it is still not clear whether the same dose of local anesthetic is similarly effective, regardless of parturient's and fetal size.

DETAILED DESCRIPTION:
Spinal block is a gold standard of cesarean section anesthesia. Two major factors contribute to its popularity: more than satisfactory level of surgical conditions and the fact that the mother is able to witness the birth of her child and both of them can benefit from skin-to-skin contact. For the procedure to proceed with patient's comfort the level of sensory block is required to be adequately high, reaching high thoracic dermatomes.

For this reason the quest for the ideal dose of local anesthetic is still ongoing. A few strategies has been proposed. Adjusting the dose to patient's size is probably the most popular. In order to minimize the risk of spinal block - related complications and maintain acceptable level of effectiveness, it was suggested that height, weight, maternal weight gain, abdominal circumference or combination of these variables may be used to calculate the appropriate spinal dose of hyperbaric bupivacaine.

In this study we will investigate whether demographic variables relate to maximal level of spinal sensory blockade when the same high dose of local anesthetic is used (close to the dose effective in 95% of cases (ED95)).

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery at term under spinal anesthesia
* American Society of Anesthesiologists (ASA) physical status <3
* BMI<40

Exclusion Criteria:

* Spinal anesthesia with the dose different than 12.5mg of hyperbaric bupivacaine
* Local anesthetic other than hyperbaric bupivacaine used
* Failed spinal anesthesia
* Poor quality of anesthetic record - required data not available

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be chosen from the cases of elective cesarean sections that took place in years 2017-2022 in Orlowski Hospital, Department of Obstetrics and Gynecology, Centre of Postgraduate Medical Education, Warsaw, Poland. Intention is to include at least 140 cases for good quality analysis
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessed variable - block level correlation coefficient | Highest level of sensory block noted from the time of spinal injection until the end of surgical procedure
  Regression and correlation analysis will be employed to assess the relation between pregnancy-related, maternal and neonatal data and the level of sensory block. For the purpose of statistical analysis the level of block will be converted into numbers for more reliable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Malec-Milewska, MD, Prof., Study Chair — Department of Anesthesia and Intensive Care, Orlowski Hospital, Warsaw
Locations (1):
- Centre of Postgraduate Medical Education,Department of Anesthesia and Intensive Care, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ozkan Seyhan T, Orhan-Sungur M, Basaran B, Savran Karadeniz M, Demircan F, Xu Z, Sessler DI. The effect of intra-abdominal pressure on sensory block level of single-shot spinal anesthesia for cesarean section: an observational study. Int J Obstet Anesth. 2015 Feb;24(1):35-40. doi: 10.1016/j.ijoa.2014.08.004. Epub 2014 Aug 27. PMID 25499016
- [Background] Bialowolska K, Horosz B, Sekowska A, Malec-Milewska M. Fixed Dose versus Height-Adjusted Conventional Dose of Intrathecal Hyperbaric Bupivacaine for Caesarean Delivery: A Prospective, Double-Blinded Randomised Trial. J Clin Med. 2020 Nov 8;9(11):3600. doi: 10.3390/jcm9113600. PMID 33171677
- [Background] Wei CN, Zhou QH, Wang LZ. Abdominal girth and vertebral column length aid in predicting intrathecal hyperbaric bupivacaine dose for elective cesarean section. Medicine (Baltimore). 2017 Aug;96(34):e7905. doi: 10.1097/MD.0000000000007905. PMID 28834913